CLINICAL TRIAL: NCT04307186
Title: Multicenter, Single-blind, Adaptive Dose Finding Study of Single Intravenous Injections of BAY 1747846 With Corresponding Blinded Read in Adult Participants With Known or Highly Suspected CNS Lesions Referred for Contrast-enhanced MRI of the CNS
Brief Title: Study to Find the Appropriate Dose of a New Gadolinium-based Contrast Agent (GBCA) for Adults Undergoing Magnetic Resonance Imaging (MRI) for Known or Highly Suspected Brain and/or Spinal Cord Conditions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20241; 2019-001560-30 (EudraCT Number)
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Central Nervous System Pathology
Keywords: CNS
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Masking Description: This is a one-way crossover study with blinded participants and blinded image readers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gadobutrol + Gadoquatrane (Experimental): Participants will receive one intravenous (IV) injection of gadobutrol 0.1 millimole(s) gadolinium/kilogram body weight (mmol Gd/kg bw) and one IV injection of Gadoquatrane (BAY1747846).
  Interventions: Drug: Gadoquatrane (BAY1747846); Drug: Gadobutrol (Gadovist/Gadavist)

INTERVENTIONS:
Drug: Gadoquatrane (BAY1747846) — Solution for IV injection, single dose
Drug: Gadobutrol (Gadovist/Gadavist) — Solution for IV injection, single dose

SUMMARY:
Researchers in this study want to find the appropriate dose of drug BAY1747846 for adults undergoing MRI for known or highly suspected brain and/or spinal cord conditions so that the image quality is similar to that of drug gadobutrol for adults undergoing MRI. MRI stands for Magnetic resonance imaging which produces body pictures created by using magnetic energy rather than x-ray energy.

Both BAY1747846 and gadobutrol are medicinal products known as gadolinium-based contrast agents (GBCA) which are used in MRI examinations to provide contrast enhancement and improve imaging performance. Gadobutrol (brand name: Gadavist, Gadovist) has been approved worldwide for the diagnosis of various disorders in adult and pediatric patients. BAY1747846 is a new GBCA under development with the goal to provide similar imaging performances in MRI. Participants in this study will receive both BAY1747846 and gadobutrol with a period of 3 - 14 days in between. A MRI examination will be performed after each injection. Participant will stay in this study for 2 - 4 weeks depending on the scheduling of the visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of signing the informed consent.
* Known or highly suspected CNS pathology (contrast-enhancing CNS lesion) referred for contrast-enhanced MRI of the CNS.
* Male and female.
* Estimated glomerular filtration rate (eGFR) value ≥ 60 mL/min/1.73m^2.

Exclusion Criteria:

* Considered clinically unstable or has a concomitant/intercurrent condition (e.g. COVID-19 infection) that would not allow participation for the full planned study period (i.e. period 1, 2 or both) in the judgement of the investigator.
* Severe cardiovascular disease.
* Patients undergoing liver transplantation.
* Any contraindication to MRI examinations.
* History of severe allergic or anaphylactic/anaphylactoid reaction to any allergen including drugs and contrast agents, foods, chemicals or other substances.
* History of allergic asthma and/ or atopic dermatitis.
* Suspected lesions or suffering from any of the following CNS diseases/lesion types as the main indication for MRI:

  * Lepto-meningeal disease (e.g. leptomeningeal carcinomatosis). Dural lesions (e.g. meningiomas) fulfilling inclusion criteria #2 are not excluded
  * Pituitary adenomas (macro and micro)
  * Tumors of the choroid plexus
  * Tumors of the pineal gland
  * Dermoid/epidermoid tumors
  * Infectious disease (e.g. brain abscess, cisticercosis, etc.)
  * Venous angiomas
  * Subacute/chronic ischemia
  * Encephalitis
  * Multiple sclerosis (acute and chronic)
  * Optic neuritis
  * Chordomas
  * Von Hippel Lindau syndrome
  * Hypertensive leukoencephalopathy.
* Receipt of any contrast agent < 72 h prior to the study MRIs, or planned receipt of any contrast agent within 72 h after the second study MRI.
* Planned or expected biopsy in the region of interest or any interventional therapeutic procedure from the first study MRI up to 24 h after the second study MRI.
* Planned or expected change in any treatment or procedure between the two study MRIs that may alter image comparability and /or chemotherapy which is changed between the two MRI procedures.
* Contraindications to the administration of gadobutrol, as specified in the local product label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- Bulgaria (3):
  - UMHAT Sveti Georgi, Plovdiv
  - Acibadem City Clinic Multiprofile Hospital for Active Treatm, Sofia
  - University Multiprofile Hosp. for Active Treat. Sveti Ivan, Sofia
- Germany (3):
  - MVZ Prof. Uhlenbrock und Partner, Dortmund, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Friedrich-Schiller-Uni. Jena, Jena, Thuringia
- Japan (8):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Himeji Medical Center, Himeji, Hyōgo
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya, Hyōgo
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - National Hospital Organization Kanmon Medical Center, Shimonoseki, Yamaguchi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 17 study centers in 4 countries between 18-Nov-2020 (first participant first visit) and 6-Sep-2022 (last participant last visit).
Pre-assignment Details: Of the 62 screened participants 5 were screening failures, resulting in 57 participants assigned to treatment who started with gadobutrol.
Groups:
- Gadobutrol + Gadoquatrane: Participants received one intravenous (IV) injection of gadobutrol 0.1 millimole(s) gadolinium/kilogram body weight (mmol Gd/kg bw) during treatment Period 1 and one IV injection of gadoquatrane (BAY1747846) 0.04 mmol Gd/kg bw during treatment Period 2.
Period: Period 1 - Gadobutrol
Arm/Group | Gadobutrol + Gadoquatrane
Started | 57
Completed | 56
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Washout 3-14 Days
Arm/Group | Gadobutrol + Gadoquatrane
Started | 56
Completed | 53
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 1
Not completed — Pre-specified withdrawal criterion met | 1
Period: Period 2 - Gadoquatrane
Arm/Group | Gadobutrol + Gadoquatrane
Started | 53
Completed | 52
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gadobutrol + Gadoquatrane
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Diagnostic Preference
Description: Overall diagnostic preference using a matched pairs approach was evaluated by 3 blinded readers using an ordinal 5-point scale (greatly prefer gadoquatrane, prefer gadoquatrane, no preference, prefer gadobutrol, greatly prefer gadobutrol). Percentage of participants and the respective Wald confidence intervals (CI) for image preference were reported for each of the 3 readers based on the 3-point preference scale (1=greatly prefer/prefer gadoquatrane, 0=no preference, -1=greatly prefer/prefer gadobutrol). If 2 or 3 readers reach the same conclusion on the recommended action (e.g. no dose adjustment needed), then this will be the recommended action taken.
Time Frame: At 5 minute post each injection
Population: Full analysis set (FAS): All participants who have completed magnetic resonance (MR) image datasets that qualify for blinded read.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gadobutrol + Gadoquatrane
Number analyzed (Participants) | 50
Percentage of participants
  Reader 1 (1) | 10 [1.68 to 18.32]
  Reader 1 (0) | 34 [20.87 to 47.13]
  Reader 1 (-1) | 56 [42.24 to 69.76]
  Reader 2 (1) | 26 [13.84 to 38.16]
  Reader 2 (0) | 42 [28.32 to 55.68]
  Reader 2 (-1) | 32 [19.07 to 44.93]
  Reader 3 (1) | 30 [17.30 to 42.70]
  Reader 3 (0) | 28 [15.55 to 40.45]
  Reader 3 (-1) | 42 [28.32 to 55.68]
Statistical Analysis 1: Comparison: Gadobutrol + Gadoquatrane; Reader 1; Test type: Other — McNemar test was used for the exploratory analysis of difference between the percentage of participants "greatly prefer/prefer gadoquatrane" and "greatly prefer/prefer gadobutrol"; p < 0.0001, McNemar — P-Value was calculated. p < 0.05 indicates a difference between the two reads; p > 0.05 indicates the observed data do not contradict equality
Statistical Analysis 2: Comparison: Gadobutrol + Gadoquatrane; Reader 2; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5775, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Gadobutrol + Gadoquatrane; Reader 3; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3173, McNemar — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Sum of Lesion Visualization Parameters on Post-contrast Images
Description: The 3 lesion visualization parameters (border delineation/degree of contrast enhancement/internal morphology) were combined by adding them up for each participant and each blinded reader, leading to only one variable on an ordinal 11-point scale (the higher values represent a better lesion visualization). Average reader was the mean of the 3 blinded readers averages of the scores per participant. Lesion border delineation: measured on a 4-point scale (1=None [no/unclear delineation of the lesion boundaries] to 4=Excellent [clear and complete delineation]). Degree of lesion contrast enhancement: measured on a 4-point scale (1=No [lesion is not enhanced] to 4=Excellent [lesion is clearly and brightly enhanced]). Lesion internal morphology: measured on a 3-point scale (1=Poor [structure and internal morphology of the lesion is poorly visible] to 3=Good [structure and internal morphology of the lesion is sufficiently visible]).
Time Frame: At 5 minute post each injection
Population: Full analysis set (FAS): All participants who have completed magnetic resonance image datasets that qualify for blinded read.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Gadobutrol Post-contrast: MR images were taken 5 min after receiving IV injection of gadobutrol.
- Gadoquatrane Post-contrast: MR images were taken 5 min after receiving IV injection of gadoquatrane.
Arm/Group | Gadobutrol Post-contrast | Gadoquatrane Post-contrast
Number analyzed (Participants) | 50 | 50
Scores on a scale
  Reader 1: number analyzed (Participants) | 49 | 49
  Reader 1 | 9.95 (1.447) | 9.67 (1.541)
  Reader 2 | 7.67 (1.292) | 7.49 (1.406)
  Reader 3: number analyzed (Participants) | 50 | 49
  Reader 3 | 9.28 (1.877) | 9.65 (1.598)
  Average reader: number analyzed (Participants) | 49 | 49
  Average reader | 9.00 (1.294) | 8.94 (1.229)
Statistical Analysis 1: Comparison: Gadobutrol Post-contrast vs Gadoquatrane Post-contrast; Average reader; Test type: Non-Inferiority — The non-inferiority of gadoquatrane versus gadobutrol was evaluated using CIs based on the t-distribution. A non-inferiority margin of 1 was used, i.e. meaning that a 95% two-sided CI for the mean difference gadoquatrane minus gadobutrol score must exclude the value -1; p < 0.0001, t-test, 1 sided — P-Value was calculated. Non-inferiority was achieved with a one-sided p-value lower than 0.025; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.24 to 0.13]

3. Secondary Outcome: Lesion Visualization Parameter Border Delineation on Pre-contrast and Combined Pre- and Post-contrast Images
Description: Lesion border delineation: up to 5 of the largest lesions were selected and scored using a 4-point scale (1=None [no/unclear delineation of the lesion boundaries] to 4=Excellent [clear and complete delineation]; the higher values represent a better lesion border delineation). Average reader was the mean of the 3 blinded readers averages of the scores per participant.
Time Frame: At pre-injection and 5 minute post each injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Gadobutrol Pre-contrast: MR images were taken before receiving IV injection of gadobutrol.
- Gadobutrol Combined Pre- and Post-contrast: Evaluation of the combined MR image sets taken before and 5 min after receiving IV injection of gadobutrol.
- Gadoquatrane Pre-contrast: MR images were taken before receiving IV injection of gadoquatrane.
- Gadoquatrane Combined Pre- and Post-contrast: Evaluation of the combined MR image sets taken before and 5 min after receiving IV injection of gadoquatrane.
Arm/Group | Gadobutrol Pre-contrast | Gadobutrol Combined Pre- and Post-contrast | Gadoquatrane Pre-contrast | Gadoquatrane Combined Pre- and Post-contrast
Number analyzed (Participants) | 50 | 50 | 50 | 50
Scores on a scale
  Reader 1: number analyzed (Participants) | 46 | 46 | 43 | 43
  Reader 1 | 1.83 (0.701) | 3.39 (0.936) | 1.88 (0.698) | 3.28 (0.970)
  Reader 2: number analyzed (Participants) | 44 | 44 | 44 | 44
  Reader 2 | 1.70 (0.509) | 2.45 (0.589) | 1.67 (0.469) | 2.39 (0.576)
  Reader 3: number analyzed (Participants) | 40 | 40 | 41 | 41
  Reader 3 | 1.98 (0.423) | 3.28 (0.751) | 1.87 (0.403) | 3.21 (0.873)
  Average reader: number analyzed (Participants) | 39 | 39 | 39 | 39
  Average reader | 1.82 (0.438) | 3.02 (0.614) | 1.81 (0.394) | 2.91 (0.609)
Statistical Analysis 1: Comparison: Gadobutrol Pre-contrast vs Gadobutrol Combined Pre- and Post-contrast; Average Reader; Test type: Other — 95% two-sided CIs based on a t-distribution for the difference of combined pre- and post-contrast minus pre-contrast scores; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [1.06 to 1.34] — Descriptive comparison of the result following gadobutrol with the result following gadoquatrane
Statistical Analysis 2: Comparison: Gadoquatrane Pre-contrast vs Gadoquatrane Combined Pre- and Post-contrast; Average Reader; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [0.94 to 1.25] — Descriptive comparison of the result following gadobutrol with the result following gadoquatrane

4. Secondary Outcome: Lesion Visualization Parameter Contrast Enhancement on Pre-contrast and Combined Pre- and Post-contrast Images
Description: Degree of lesion contrast enhancement: up to the 5 largest lesions were selected and scored using a 4-point scale (1=No [lesion is not enhanced] to 4=Excellent [lesion is clearly and brightly enhanced]; the higher values represent a better degree of lesion contrast enhancement). Average reader was the mean of the 3 blinded readers averages of the scores per participant.
Time Frame: At pre-injection and 5 minute post each injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadobutrol Pre-contrast | Gadobutrol Combined Pre- and Post-contrast | Gadoquatrane Pre-contrast | Gadoquatrane Combined Pre- and Post-contrast
Number analyzed (Participants) | 50 | 50 | 50 | 50
Scores on a scale
  Reader 1: number analyzed (Participants) | 46 | 46 | 43 | 43
  Reader 1 | 1.00 (0.000) | 3.24 (0.917) | 1.00 (0.000) | 3.20 (0.825)
  Reader 2: number analyzed (Participants) | 44 | 44 | 44 | 44
  Reader 2 | 1.00 (0.000) | 2.50 (0.629) | 1.00 (0.000) | 2.57 (0.587)
  Reader 3: number analyzed (Participants) | 40 | 40 | 41 | 41
  Reader 3 | 1.00 (0.000) | 3.55 (0.904) | 0.99 (0.078) | 3.49 (0.925)
  Average Reader: number analyzed (Participants) | 39 | 39 | 39 | 39
  Average Reader | 1.00 (0.000) | 3.07 (0.638) | 1.00 (0.027) | 3.05 (0.600)
Statistical Analysis 1: Comparison: Gadobutrol Pre-contrast vs Gadobutrol Combined Pre- and Post-contrast; Average Reader; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.07, 95% CI 2-sided [1.87 to 2.28] — Descriptive comparison of the result following gadobutrol with the result following gadoquatrane
Statistical Analysis 2: Comparison: Gadoquatrane Pre-contrast vs Gadoquatrane Combined Pre- and Post-contrast; Average Reader; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.06, 95% CI 2-sided [1.86 to 2.25] — Descriptive comparison of the result following gadobutrol with the result following gadoquatrane

5. Secondary Outcome: Lesion Visualization Parameter Internal Morphology on Pre-contrast and Combined Pre- and Post-contrast Images
Description: Lesion internal morphology: up to 5 of the largest lesions were selected and scored using a 3-point scale (1=Poor [structure and internal morphology of the lesion is poorly visible] to 3=Good [structure and internal morphology of the lesion is sufficiently visible]; the higher values represent a better lesion internal morphology). Average reader was the mean of the 3 blinded readers averages of the scores per participant.
Time Frame: At pre-injection and 5 minute post each injection
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadobutrol Pre-contrast | Gadobutrol Combined Pre- and Post-contrast | Gadoquatrane Pre-contrast | Gadoquatrane Combined Pre- and Post-contrast
Number analyzed (Participants) | 50 | 50 | 50 | 50
Scores on a scale
  Reader 1: number analyzed (Participants) | 46 | 46 | 43 | 43
  Reader 1 | 1.27 (0.444) | 2.62 (0.693) | 1.40 (0.484) | 2.58 (0.655)
  Reader 2: number analyzed (Participants) | 44 | 44 | 44 | 44
  Reader 2 | 1.05 (0.185) | 2.13 (0.598) | 1.05 (0.211) | 2.11 (0.689)
  Reader 3: number analyzed (Participants) | 40 | 40 | 41 | 41
  Reader 3 | 1.05 (0.221) | 2.45 (0.677) | 1.04 (0.234) | 2.44 (0.673)
  Average Reader: number analyzed (Participants) | 39 | 39 | 39 | 39
  Average Reader | 1.13 (0.194) | 2.39 (0.493) | 1.16 (0.218) | 2.35 (0.500)
Statistical Analysis 1: Comparison: Gadobutrol Pre-contrast vs Gadobutrol Combined Pre- and Post-contrast; Average Reader; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.27, 95% CI 2-sided [1.11 to 1.43] — Descriptive comparison of the result following gadobutrol with the result following gadoquatrane
Statistical Analysis 2: Comparison: Gadoquatrane Pre-contrast vs Gadoquatrane Combined Pre- and Post-contrast; Average Reader; Test type: Other — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [1.05 to 1.32] — Descriptive comparison of the result following gadobutrol with the result following gadoquatrane

6. Secondary Outcome: Number of Lesions on Pre-contrast and Combined Pre- and Post-contrast Images
Description: The 3 blinded readers recorded the total number of lesions for each pre-contrast and combined pre- and post-contrast magnetic resonance image set separately. The numbers of participants by number of detected lesions were reported.
Time Frame: At pre-injection and 5 minute post injection
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Gadobutrol Pre-contrast: Magnetic resonance (MR) images were taken before receiving IV injection of gadobutrol.
Arm/Group | Gadobutrol Pre-contrast | Gadobutrol Combined Pre- and Post-contrast | Gadoquatrane Pre-contrast | Gadoquatrane Combined Pre- and Post-contrast
Number analyzed (Participants) | 50 | 50 | 50 | 50
Participants
  Reader 1 (Nr. of lesions=0) | 4 | 1 | 7 | 1
  Reader 1 (Nr. of lesions=1) | 43 | 40 | 40 | 41
  Reader 1 (Nr. of lesions=2) | 3 | 7 | 1 | 6
  Reader 1 (Nr. of lesions=3) | 0 | 2 | 2 | 2
  Reader 2 (Nr. of lesions=0): number analyzed (Participants) | 48 | 49 | 49 | 49
  Reader 2 (Nr. of lesions=0) | 4 | 0 | 5 | 0
  Reader 2 (Nr. of lesions=1): number analyzed (Participants) | 48 | 49 | 49 | 49
  Reader 2 (Nr. of lesions=1) | 42 | 43 | 42 | 43
  Reader 2 (Nr. of lesions=2): number analyzed (Participants) | 48 | 49 | 49 | 49
  Reader 2 (Nr. of lesions=2) | 0 | 3 | 0 | 3
  Reader 2 (Nr. of lesions=3): number analyzed (Participants) | 48 | 49 | 49 | 49
  Reader 2 (Nr. of lesions=3) | 2 | 3 | 2 | 3
  Reader 3 (Nr. of lesions=0) | 10 | 1 | 9 | 1
  Reader 3 (Nr. of lesions=1) | 40 | 41 | 40 | 42
  Reader 3 (Nr. of lesions=2) | 0 | 7 | 1 | 4
  Reader 3 (Nr. of lesions=3) | 0 | 1 | 0 | 1
  Reader 3 (Nr. of lesions=4) | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events tables: up to the 24 h ± 4 h follow-up time point following Gadobutrol or Gadoquatrane injection. All-cause mortality table: after signing informed consent up to the last contact per participant, up to 36 days.
Groups:
- Gadobutrol: Participants received one intravenous (IV) injection of gadobutrol 0.1 millimole(s) gadolinium/kilogram body weight (mmol Gd/kg bw) during treatment Period 1.
- Gadoquatrane: Participants received one IV injection of gadoquatrane (BAY1747846) 0.04 mmol Gd/kg bw during treatment Period 2.
Arm/Group | Gadobutrol | Gadoquatrane
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/52
Other Adverse Events (participants affected / at risk) | 3/57 | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol (N=57) | Gadoquatrane (N=52)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A written manuscript of any oral/written publication relating to the trial, the investigational medicinal products or the results shall be submitted to Bayer for review at least 60 days before the planned filing or presentation of the publication. If Bayer does not confirm receipt of the intended publication within 45 days, Bayer must be informed again of the intended publication date. If Bayer does not comment on the publication within the 60-day period, the publication is free to be published.

DOCUMENTS (2):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT04307186/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04307186/SAP_001.pdf